CLINICAL TRIAL: NCT05593120
Title: Evaluation of Health Economics for Noninvasive Coronary Fractional Flow Reserve Measurement Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Raysight Intelligent Medical Technology Co., Ltd. (Industry)
Collaborators: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Health Economics
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CT-FFR: All patients will be assessed and managed according to the results of CT-FFR test, assuming they have no prespecified contraindications to CT coronary angiography. The result of the CT-FFR will be conveyed to the supervising physician within 24 hours and will be used to determine the subsequent management plan.
  Interventions: Diagnostic Test: CT-FFR
- Routine care: All patients will be assessed and managed exactly as they are usually treated by the investigator and the institution's heart team according to routine practice in Wuhan Asia Heart Hospital.
  Interventions: Diagnostic Test: Routine care

INTERVENTIONS:
Diagnostic Test: CT-FFR — In the test group all patients who are eligible for CTA will undergo CTA as their default test. Those patients with any coronary stenosis 30%-90% data in at least one major epicardial vessel will be referred for CT-FFR. In patients in whom CT-FFR analysis is performed, FFR will be derived for all vessels. CT-FFR will be evaluated in a blinded fashion with a "Coarse-to-Fine Subpixel" algorithm for lumen contour. The data derived from this test will determine their management strategy.
  Groups: CT-FFR
Diagnostic Test: Routine care — All patients in the routine care group will be assessed according to their current conventional pathways that are based upon routine practice in Wuhan Asia Heart Hospital. The trial will encourage the routine and standard assessment and management of all patients (anticipated outcomes include ETT, stress echo, stress MR, nuclear perfusion, CTA, CT calcium, invasive CA, reassurance).
  Groups: Routine care

SUMMARY:
To determine whether, in a Chinese population of patients presenting to Wuhan Asia Heart Hospital, Fractional Flow Reserve Derived from Coronary Computed Tomography Angiography (CT-FFR) as a default test is noninferior in terms of total costs when compared to routine clinical pathway recommended by the investigator and the institution's heart team.

DETAILED DESCRIPTION:
The 2021 ACC/AHA Guidelines now highlight use of CT-FFR as a front-line pathway to help in "the diagnosis of vessel-specific ischemia and to guide decision-making regarding the use of coronary revascularization". Previous observational PLATFORM study, which compared the use of CT-FFR with standard assessment of patients with stable chest pain enrolled from 11 European sites, demonstrated that management based on CT-FFR was both safe and associated with a significantly lower frequency of invasive angiograms demonstrating no significant coronary artery disease (CAD). Furthermore, the CT-FFR strategy appeared to be economically attractive in this observational study, and was supported by the 2016 National Institute for Health and Care Excellence (NICE) guidance. In contrast, the FORECAST randomized trial included 1400 patients with stable chest pain from 11 centres in the UK, and the results showed that a strategy of CCTA with selective CT-FFR in patients with stable angina did not differ significantly from standard clinical care pathways in cost or clinical outcomes, but did reduce the use of invasive coronary angiography. As abovementioned, the population enrolled in the previous studies were from different western countries, and the cost analysis results of CT-FFR application in different countries are diverse in terms of health care economics.

To date, however, the cost-effectiveness and clinical safety impact of using CT-FFR instead of other tests in the initial evaluation of patients with suspected coronary artery disease has not been tested in a prospective clinical trial in China.

The OVERALL OBJECTVE of this prospective, observational study is to compare resource utilization, time-effectiveness and clinical safety in subjects with suspected CAD receiving standard practice evaluation and treatment versus subjects receiving CT-FFR-guided evaluation and treatment in order to further inform patients, health care providers, and other stakeholders about which technologies are most cost-effective and efficient in the diagnosis of CAD. The hypothesis this CERTAIN trial is that CT-FFR would be associated with (1) lower overall costs; (2) shorter time period between initial consultation and definitive management plan; (3) better patient experience.

The 2 strategies for the CERTAIN trial are:

[A] TEST GROUP: All patients will be assessed and managed according to the results of CT-FFR test, assuming they have no prespecified contraindications to CT coronary angiography. The result of the CT-FFR will be conveyed to the supervising physician within 24 hours and will be used to determine the subsequent management plan.

[B] REFERENCE GROUP: All patients will be assessed and managed exactly as they are usually treated by the investigator and the institution's heart team according to standard practice in Wuhan Asia Heart Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Providing written informed consent
* No contraindication to CTA
* At least 1 lesion with a percent diameter stenosis (DS%) 30%-90% in a coronary artery with a ≥2.0 mm reference vessel diameter diagnosed on coronary CTA

Exclusion Criteria:

* Acute coronary syndrome or myocardial infarction requiring urgent revascularization
* Prior PCI or CABG surgery
* Allergic to contrast
* BMI>35 at the time of coronary CTA
* Advanced renal impairment
* Significant valve disease (severe aortic stenosis or regurgitation; severe mitral regurgitation)
* Life expectancy <12 months
* Repeated enrollment
* Any other factors that the researchers consider not suitable for inclusion or completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with at least 1 lesion with a percent diameter stenosis (DS%) 30%-90% in a coronary artery with a ≥2.0 mm reference vessel diameter diagnosed on coronary CTA, suspected CAD
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Resource utilisation | 6 months
  To determine whether, in a Chinese population of patients presenting to Wuhan Asia Heart Hospital, CT-FFR as a default test is noninferior in terms of total costs when compared to routine clinical pathway recommended by the investigator and the institution's heart team. Comparison of resource utilization between two groups at 180 days (+30/-15 days).

SECONDARY OUTCOMES:
time period between initial consultation and definitive management plan | 6 months
  Comparison of time period between initial consultation and definitive management plan between two groups during 180 days (+30/-15 days).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Ma, Principal Investigator — Wuhan Asia Heart Hospital
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, Hubei, China